CLINICAL TRIAL: NCT00894920
Title: Biotin Status in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 3114301; R01DK079892-01 (NIH); 107068
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Biotin Deficiency
Keywords: biotin; deficiency; pregnancy; lymphocyte propionyl-CoA carboxylase
MeSH Terms: conditions — Biotin deficiency | interventions — Biotin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: biotin
- biotin (Active Comparator)
  Interventions: Dietary Supplement: biotin

INTERVENTIONS:
Dietary Supplement: biotin — capsule approximately 30 mcg daily 21 days
  Arms: placebo
Dietary Supplement: biotin — capsule 300 mcg daily 21 days
  Arms: biotin

SUMMARY:
The purpose of this study is to estimate the number of pregnant women who, during pregnancy, have low levels of the vitamin biotin. The hypothesis of this study is that a large number of pregnant women will have low biotin levels. This information will be used to later determine if low biotin levels during pregnancy cause certain birth defects.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40
* in early pregnancy (less than 15 weeks gestation)
* under care of physician
* normal pregnancy
* taking prenatal vitamin with less than 30 mcg biotin

Exclusion Criteria:

* prenatal vitamin with greater than 30 mcg biotin
* antibiotic use
* known renal disease
* drug, alcohol abuse
* gastric bypass
* daily diet high in biotin
* use of certain meal replacement products high in biotin
* previous history of children with birth defects

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2009-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Lymphocyte propionyl-CoA carboxylase (PCC) activities | 2-3 months

SECONDARY OUTCOMES:
Urinary biotin excretion | 2-3 months
Urinary 3-hydroxyisovaleric acid (3HIA) excretion | 2-3 months
Other biotin-related indicators in urine and blood | 2-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Mock, MD,PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States